CLINICAL TRIAL: NCT03091660
Title: S1602, A Phase III Randomized Trial to Evaluate the Influence of BCG Strain Differences and T Cell Priming With Intradermal BCG Before Intravesical Therapy for BCG-Naive High-Grade Non-muscle Invasive Bladder Cancer
Brief Title: S1602: Different Strains of BCG With or Without Vaccine in High Grade Non- Muscle Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1602; NCI-2016-00451 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1602 (Other: SWOG); S1602 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stage 0 Bladder Urothelial Carcinoma; Stage 0is Bladder Urothelial Carcinoma; Stage I Bladder Urothelial Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (BCG solution) (Active Comparator): INDUCTION: Patients receive TICE BCG solution intravesically once a week for 6 weeks. MAINTENANCE: Patients receive TICE BCG solution once a week for 3 consecutive weeks at months 3, 6, 12, 18, 24, 30, and 36 for up to 7 doses.
  Interventions: Biological: BCG Solution; Other: Laboratory Biomarker Analysis
- Arm II (Tokyo-172 strain BCG solution) (Experimental): INDUCTION: Patients receive Tokyo-172 strain BCG solution intravesically once a week for 6 weeks. MAINTENANCE: Patients receive Tokyo-172 strain BCG solution once a week for 3 consecutive weeks at months 3, 6, 12, 18, 24, 30, and 36 for up to 7 doses.
  Interventions: Biological: BCG Tokyo-172 Strain Solution; Other: Laboratory Biomarker Analysis
- Arm III (Tokyo-172 strain BCG solution with priming) (Experimental): PRIME: Patients receive Tokyo-172 strain BCG vaccine once ID. INDUCTION: Within 21 days, patients receive Tokyo-172 strain BCG solution as in Arm II. MAINTENANCE: Patients receive Tokyo-172 strain BCG solution as in Arm II.
  Interventions: Biological: BCG Tokyo-172 Strain Solution; Biological: BCG Tokyo-172 Strain Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: BCG Solution — Given intravesically
  Other Names: Bacillus Calmette-Guerin Solution; TICE BCG Solution
  Arms: Arm I (BCG solution)
Biological: BCG Tokyo-172 Strain Solution — Given intravesically
  Other Names: Bacillus Calmette-Guerin Tokyo-172 Strain Solution; Immunobladder
  Arms: Arm II (Tokyo-172 strain BCG solution); Arm III (Tokyo-172 strain BCG solution with priming)
Biological: BCG Tokyo-172 Strain Vaccine — Given ID
  Other Names: Bacillus Calmette-Guerin Tokyo-172 Strain Vaccine
  Arms: Arm III (Tokyo-172 strain BCG solution with priming)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase III trial studies Tokyo-172 strain bacillus Calmette-Guerin (BCG) solution with or without a vaccination using Tokyo-172 strain BCG to see how well it works compared with TICE BCG solution in treating patients with bladder cancer that has not spread to muscle. BCG is a non-infectious bacteria that when instilled into the bladder may stimulate the immune system to fight bladder cancer. Giving different versions of BCG with vaccine therapy may prevent bladder cancer from returning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare whether time to high grade recurrence (TTHGR) for patients with BCG-naïve, non-muscle invasive bladder cancer (NMIBC) receiving Tokyo-172 BCG strain (Arm II) is non-inferior to patients receiving TICE BCG strain (Arm I).

II. To test whether TTHGR for patients with BCG-naïve, NMIBC receiving intradermal Tokyo-172 BCG vaccination followed by intravesical Tokyo-172 BCG instillation (Arm III) is superior to patients receiving intravesical Tokyo-172BCG instillation without prior intradermal BCG vaccination (Arm II).

SECONDARY OBJECTIVES:

I. To compare time to recurrence (TTR) with any-grade (AG) bladder cancer between patients receiving Tokyo-172 versus TICE BCG strain.

II. To compare TTR with AG bladder cancer between patients receiving intradermal + intravesical versus intravesical only Tokyo-172 BCG.

III. To compare progression-free survival (PFS) between patients receiving Tokyo-172 versus TICE BCG strain.

IV. To compare PFS between patients receiving intradermal + intravesical versus intravesical only Tokyo-172 BCG.

V. To compare 6-month complete response in patients with carcinoma in situ (CIS) with or without Ta or T1 cancer present at baseline receiving Tokyo-172 versus TICE BCG strain.

VI. To compare 6-month complete response in patients with CIS with or without Ta or T1 cancer present at baseline receiving intradermal + intravesical versus intravesical only Tokyo-172 BCG.

TERTIARY OBJECTIVES:

I. To test the hypothesis that purified protein derivative (PPD) test conversion (positive PPD at 3 or 6 months) following BCG immunotherapy will predict time to high grade recurrence (TTHGR).

II. To test the hypothesis that urinary cytokine levels following BCG immunotherapy will predict time to high grade recurrence (TTHGR).

III. To test the hypothesis that tumor neoantigen burden and T lymphocyte infiltration are associated with BCG response.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I:

INDUCTION: Patients receive TICE BCG solution intravesically once a week for 6 weeks.

MAINTENANCE: Patients receive TICE BCG solution once a week for 3 consecutive weeks at months 3, 6, 12, 18, 24, 30, and 36 for up to 7 doses.

ARM II:

INDUCTION: Patients receive Tokyo-172 strain BCG solution intravesically once a week for 6 weeks.

MAINTENANCE: Patients receive Tokyo-172 strain BCG solution once a week for 3 consecutive weeks at months 3, 6, 12, 18, 24, 30, and 36 for up to 7 doses.

ARM III:

PRIME: Patients receive Tokyo-172 strain BCG vaccine once intradermally (ID).

INDUCTION: Within 21 days, patients receive Tokyo-172 strain BCG solution as in Arm II.

MAINTENANCE: Patients receive Tokyo-172 strain BCG solution as in Arm II.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven Ta, carcinoma in situ (CIS) or T1 stage urothelial cell carcinoma of the bladder within 90 days of registration
* Patients must have had all grossly visible papillary tumors removed within 30 days prior to registration or cystoscopy confirming no grossly visible papillary tumors within 30 days prior to registration
* Patients with T1 disease must have cross-sectional imaging of abdomen/pelvis demonstrating no evidence of metastatic disease (magnetic resonance imaging [MRI] or computed tomography [CT] scan) within 90 days prior to registration; patients with T1 disease must have re-resection confirming =< T1 disease within 90 days prior to registration
* Patients must have high-grade bladder cancer as defined by 2004 World Health Organization (WHO)/International Society of Urological Pathology (ISUP) classification
* Patients must not have pure squamous cell carcinoma or adenocarcinoma
* Patients' disease must not have micropapillary components
* Patients must have no evidence of upper tract (renal pelvis or ureters) cancer confirmed by one of the following tests performed within 90 days prior to registration: CT urogram, intravenous pyelogram, magnetic resonance (MR) urogram, or retrograde pyelograms
* Patients must not have nodal involvement or metastatic disease
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years; patients with localized prostate cancer who are being followed by an active surveillance program are also eligible
* Patients must have a Zubrod performance status of 0-2
* Patients must not have received prior intravesical BCG
* Patients must not have known history of tuberculosis
* Patients must be PPD negative within 90 days prior to registration; PPD negativity is defined as < 10 mm diameter induration (palpable, raised hardened area) in the volar forearm at 48-72 hours following injection with standard tuberculin dose (5 units, 0.1 ml)
* Patients must be >= 18 years of age
* Patients must not be taking oral glucocorticoids at the time of registration
* Patients must not be planning to receive concomitant biologic therapy, hormonal therapy, chemotherapy, surgery, or other cancer therapy while on study
* Prestudy history and physical must be obtained within 90days prior to registration
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must be offered the opportunity to participate in specimen banking for future studies to include translational medicine studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
TTHGR for Arm I compared to Arm II | Time from randomization to first high grade recurrence assessed up to 5 years
  Time to High Grade Recurrence
TTHGR for Arm II compared to Arm III | Time from randomization to first high grade recurrence assessed up to 5 years
  Time to High Grade Recurrence

SECONDARY OUTCOMES:
Disease free rates | At 6 months
  Rates of patients who are disease free at six months versus not

CONTACTS AND LOCATIONS:
Overall Officials: Robert Svatek, Principal Investigator — SWOG Cancer Research Network
Locations (174):
- United States (174):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Island Urology-Hilo, Hilo, Hawaii
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
https://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Derived] Svatek RS, Tangen C, Delacroix S, Lowrance W, Lerner SP. Background and Update for S1602 "A Phase III Randomized Trial to Evaluate the Influence of BCG Strain Differences and T Cell Priming with Intradermal BCG Before Intravesical Therapy for BCG-naive High-grade Non-muscle-invasive Bladder Cancer. Eur Urol Focus. 2018 Jul;4(4):522-524. doi: 10.1016/j.euf.2018.08.015. Epub 2018 Sep 6. PMID 30197040